CLINICAL TRIAL: NCT03098732
Title: A Prospective International Multicentre Randomised Controlled Single Blind Clinical Investigation of Magnetically Enhanced Diffusion for Acute Ischaemic Stroke (MEDIS)
Brief Title: Magnetically Enhanced Diffusion for Acute Ischaemic Stroke (MEDIS) Trial
Acronym: MEDIS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategic hold
Sponsor: Pulse Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEDIS-INT16-002
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Infarction, Middle Cerebral Artery; Strokes Thrombotic; Neurologic Disorder; Cerebrovascular Disorders; Intracranial Embolism and Thrombosis
Keywords: Stroke; Ischemic; Tissue Plasminogen Activator; Thrombolysis; Vascular Diseases; Cerebrovascular Disorders; Fibrinolytic Agents; Plasminogen
MeSH Terms: conditions — Stroke; Ischemic Stroke; Infarction, Middle Cerebral Artery; Thrombotic Stroke; Nervous System Diseases; Cerebrovascular Disorders; Intracranial Embolism and Thrombosis; Ischemia; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to receive active treatment or sham. Enrollment will be stratified based upon age (<75 or >/=75) and location of the occlusion (M1, M2 or carotid terminus.)
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be masked with regard to treatment group. Imaging data will be evaluated by independent readers (2) blinded to treatment allocation.
  Neurological outcomes will be measured at the 90 Day visit by evaluators blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Magnetically Enhanced Diffusion (MED) (Experimental): The Experimental Treatment will receive the complete MED System Procedure consisting of MED MicroBeads and the MED Workstation magnet procedure for 60 minutes in addition to IV tissue plasminogen activator (tPA or Alteplase).
  Interventions: Device: Magnetically Enhanced Diffusion (MED)
- MED Workstation Magnet Sham Control (Sham Comparator): The MED Workstation Magnet Sham Comparator will not receive MED MicroBeads while the MED Workstation Magnet will be activated as a Sham control for 60 minutes in addition to IV tissue plasminogen activator (tPA or Alteplase).
  Interventions: Device: MED Workstation Magnet Sham Control

INTERVENTIONS:
Device: Magnetically Enhanced Diffusion (MED) — Treatment of Acute Ischemic Stroke with IV tPA and the adjunctive Magnetically Enhanced Diffusion (MED) System Procedure.
  Other Names: MED Workstation; MED MicroBeads
  Arms: Magnetically Enhanced Diffusion (MED)
Device: MED Workstation Magnet Sham Control — Treatment of Acute Ischemic Stroke with IV tPA and Sham use of the MED Workstation only, without the injection of MED MicroBeads.
  Arms: MED Workstation Magnet Sham Control

SUMMARY:
The objective of the MEDIS study is to determine if subjects experiencing an Acute Ischaemic Stroke due to large vessel occlusion, treated with IV tPA combined with the MED procedure have a greater likelihood of recanalisation 30-90 minutes after the completion of tPA infusion than subjects treated with IV tPA (plus sham device). Safety of the MED System Procedure will be evaluated by the incidence of symptomatic PH-2 haemorrhagic transformation within 24 hours following the procedure. Lastly, a health economics study will be conducted to estimate health care costs for each treatment.

DETAILED DESCRIPTION:
The study is a global, multicentre prospective, randomised, single blind, blinded endpoint study comparing rates of early recanalisation (defined by mAOL) in Acute Ischaemic Stroke (AIS) subjects with visible occlusion who are treated with either IV tPA plus sham device or IV tPA in combination with the MED System procedure.

The study population will be randomised 1:1 into two arms:

* A Sham Control Group (SCG) and an
* Experimental Treatment Group (ETG).

The ETG will receive IV tPA and the complete MED System procedure consisting of MED MicroBeads and the MED Workstation magnet procedure. The SCG will not receive MED MicroBeads while the MED Workstation will be activated as a Sham control. Subjects will be blinded to treatment arm. Stratification will be performed based upon baseline age and location of the occlusion (Middle Cerebral Artery segments M1, M2, or Carotid Terminus).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <85
2. Clinical signs consistent with acute ischaemic stroke
3. Prestroke functional independence (prestroke Modified Rankin Score ≤2)
4. NIHSS 4-25 at the time of randomisation
5. Initiation of IV tPA (alteplase or tissue Plasminogen Activator) within the locally approved time window from stroke symptom onset (onset time is defined as the last time when the subject was witnessed to be at baseline).
6. Arterial Occlusive Lesion (mAOL ≤1) in the M1 or M2 segments of the MCA (Middle Cerebral Artery) or carotid terminus confirmed by CT angiography.
7. Subject is able to start the MED procedure within 15 +10 minutes) from the t-PA IV infusion, and complete 60+15 minutes of MED procedure treatment.
8. Subject or subject's legally authorised representative has signed and dated an Informed Consent Form according to country regulations, ethics committee, and/or Institutional Review Board requirements.
9. It is the enrolling Investigator's or designee's opinion based upon the knowledge of the Subject's condition as well as the features of the MED device, that the Subject is an appropriate candidate for stroke management utilizing MED.

Exclusion Criteria:

1. The subject is likely to receive intra-arterial (IA) intervention.
2. Standard exclusions for thrombolysis according to the approved label and local institutional protocols.
3. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
4. Rapid neurological improvement prior to study randomisation suggesting resolution of the occlusion.
5. Known hyper-sensitivity to radiographic contrast agents.
6. Known hyper-sensitivity to iron-based agents or polyethylene glycol.
7. Known or suspected symptomatic haemosiderosis or haemochromatosis.
8. Has a previous or existing cardiovascular condition resulting in history of heart block, tachybrady syndrome, symptomatic postural hypotension requiring medical intervention.
9. Current participation or participation in the last 4 weeks in another investigational drug or device treatment study.
10. Life expectancy of less than 90 days due to other medical condition.
11. Subject with a pre-existing neurological or psychiatric disease that would confound the neurological and functional evaluations.
12. Subject has contraindications to Magnetic Resonance Imaging (MR; examples include, but are not limited to, an implantable cardioverter defibrillator, pacemaker, clipped or coiled aneurysm, neurostimulator).
13. Subject has recently (within 30 days) received iron replacement therapy or iron based MR contrast.
14. Subject has known or suspected liver disease, including hepatitis and/or cirrhosis.

Imaging Exclusion Criteria:

1. Computed tomography (CT) or MRI evidence of haemorrhage on presentation.
2. Exclusion: Large core of ischemia defined as NCCT ASPECTS 4 or less.
3. CT or MRI evidence of mass effect or intra-cranial tumour (except small meningioma).
4. CTA or MRA (CT or MR Angiography) evidence of carotid dissection or complete cervical carotid occlusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Performance: Early Recanalisation 60 +/- 30 minutes after IV tPA completion | 60 +/- 30 minutes after completion of IV tPA administration.
  Early recanalisation (Arterial Occlusive Lesion [mAOL] score) assessed from a blinded evaluation of Computed Tomographic Angiography (CTA) imaging of the primary lesion 60+/- 30 minutes after completion of tPA infusion. An ordinal shift analysis of the mAOL score distribution between the Sham Control and MED System Procedure arms will be conducted.
Primary Safety: Incidence of Symptomatic Type 2 Parenchymal (PH-2) Haemorrhagic Transformation | 24 ± 6 Hours after treatment
  Incidence of symptomatic PH-2 haemorrhagic transformation at 24 ± 6 hours post randomisation as determined by NCCT combined with a neurological deterioration that includes an increase of 4 points or more on the NIHSS from baseline or the lowest NIHSS value between baseline and 24 hours, or leading to death.

SECONDARY OUTCOMES:
Secondary Clinical Performance Endpoint: Neurological outcome mRS at 90 days | 90 days after randomisation
  Neurological outcome as defined by modified Rankin score (mRS) at 90 days.
Secondary Technical Clinical Performance Endpoint: Cerebral Infarct volume at 24 Hours | 24 ± 6 hours after randomisation
  Volume of cerebral infarction as measured by Non-Contrast Computed Tomography (NCCT) at 24 ± 6 hours post randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Muir, MBChB, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Countess of Chester Hospital NHS Foundation Trust, Chester

IPD SHARING:
Plan to Share IPD: No